CLINICAL TRIAL: NCT00986128
Title: A Comparative Study of the Steady State Pharmacokinetics of Lithium Before and During Multiple Oral Daily Topiramate (RWJ-17021) Dosing in Patients With Bipolar Disorders
Brief Title: A Pharmacokinetic Study of Lithium Before and During Topiramate Dosing in Bipolar Disorder Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Senior Director, Clinical Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002860
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Bipolar Disorder
Keywords: Topiramate; Lithium; Bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Topiramate

ARMS (2):
- 001 (Experimental)
  Interventions: Drug: topiramate
- 002 (Experimental)
  Interventions: Drug: topiramate

INTERVENTIONS:
Drug: topiramate — 100 mg tablet twice daily for 3 weeks
  Arms: 001
Drug: topiramate — One 100 mg and one 200 mg tablet twice daily for 3 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to determine the initial (after 1-week of maintenance dosing) and extended (after 3-weeks of maintenance dosing) effect of topiramate, at doses up to 600 mg/day, on the steady-state pharmacokinetics (absorption, distribution and excretion of the drug by the body) of lithium carbonate in patients with bipolar disorders.

DETAILED DESCRIPTION:
This was an open-label (both the investigator and the patient knew the identity of the study drug), sequential treatment, multicenter study evaluating the interaction of topiramate and lithium in patients with bipolar disorders. The study population included 24 patients (12 patients per group) with complete data considered adequate to fully evaluate the extent of the effect of topiramate on lithium pharmacokinetics (PK). The study consisted of a screening phase, during which patients were maintained on a stable dose of an immediate release lithium carbonate formulation administered every 12 hours, for a minimum of 2 weeks prior to the start of the study, and an open-label treatment phase consisting of a topiramate titration phase and a lithium and topiramate maintenance phase, and 3 PK sampling periods (days when multiple blood and urine samples are taken to estimate the amount of topiramate and /or lithium in the patients blood or urine). The duration of all of the periods were determined by the investigator. Patients were sequestered for 48 hours for each of the 3 PK sampling periods. At each sampling period, blood and urine samples were collected for laboratory safety analyses at the same designated serial sampling times and collection intervals as for PK sampling. All doses of study medication were administered every 12 hours. During PK sampling Period 1, patients were maintained on their respective morning and evening doses of lithium carbonate. Serial blood and urine samples were collected through 12 hours postdose for estimation of lithium serum and urine concentrations. Patients continued their lithium regimens and subsequently were initiated on topiramate and assigned to either the low-dose Group 1 (200 mg/day) or high-dose Group 2 (up to 600 mg/day). During the topiramate titration phase, the initial dose of topiramate was 25 mg/day and was titrated upward until the target dose of 200 mg/day was reached (Group 1) or the target dose of 600 mg/day (or maximum tolerated dose greater than 200 mg/day) was reached (Group 2). Topiramate dose titration was conducted on study Days 2, 4, and 7 for Group 1 and on Days 2, 7, 12, 17, 22, and 27 for Group 2. Once the maximum dose of topiramate was reached, the lithium and topiramate maintenance phase began and lasted for 3 weeks, during which the patients were maintained on a constant daily dose of topiramate and lithium carbonate. One week after beginning maintenance on topiramate and lithium carbonate, patients entered PK sampling Period 2 of the study, during which serial blood and urine samples were collected through 12 hours postdose for estimation of lithium serum and urine concentrations and for estimation of topiramate plasma concentrations. At the end of the 3 weeks of lithium and topiramate maintenance, patients entered PK sampling Period 3 of the study, during which serial blood and urine samples were collected through 12 hours postdose for estimation of lithium serum and urine concentrations and for estimation of topiramate plasma concentrations. Throughout the topiramate titration phase and the lithium and topiramate maintenance phase, serum trough concentrations of lithium (the amount of lithium in the patients blood immediately before their next dose) were determined prior to the morning dose every 3 days, beginning on Day 3 of the topiramate titration phase. Patients are maintained on a stable dose of an immediate release lithium carbonate formulation for 2 weeks prior to study start. In the titration phase, topiramate given every 12 hours starting at 25 mg/day. Patients are titrated to target doses of 200 mg/day (low-dose group) over a period of up to 10 days, or 600 mg/day (high-dose group) over a period of up to 30 days. The lithium and topiramate maintenance phase lasts for an additional 3 weeks after target doses are reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting DSM-IV criteria for either Bipolar I, Bipolar II, Cyclothymic Disorder, or Bipolar Disorder NOS
* Patients on monotherapy treatment with lithium carbonate at steady state level for a minimum of two weeks prior to study treatment assignment
* Women are postmenopausal for at least 1 year, or surgically incapable of childbearing, or practicing an acceptable method of birth control (hormonal contraception, intrauterine device, or barrier with spermicide were acceptable) and not pregnant at baseline

Exclusion Criteria:

* Patients with a history of an acquired or hereditary neurologic disease, e.g., epilepsy or significant brain trauma
* Patients on depot medications, including but not limited to haloperidol, decanoate and Depo-Provera
* Patients who had taken acetazolamide, zonisamide, triamterene, dichlorphenamide, chronic antacids, or calcium supplements, or any medication associated with nephrolithiasis (kidney stone formation) in the month prior to beginning topiramate titration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2001-03; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential pharmacokinetic interaction between topiramate and lithium in patients with bipolar disorders | In each sampling period, blood (lithium and topiramate concentrations) is collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-morning dose, and urine (lithium concentration) was collected at 0-2, 2-4, 4-8, and 8-12 hours postdose

SECONDARY OUTCOMES:
No Secondary Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A comparative study of the steady-state pharmacokinetics of lithium before and during multiple oral daily topiramate (RWJ-17021) dosing in patients with bipolar disorders — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=494&filename=CR002860_CSR.pdf